CLINICAL TRIAL: NCT07147452
Title: Sentinel Lymph Node Detection in Gastric Cancer Using a Dual Tracer (Superparamagnetic Iron Oxide and Methylene Blue): A Prospective Study With Histological and OSNA Validation
Acronym: SLN_GC_SPIO
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital del SAS de Jerez (Other)
Collaborators: Sysmex España (Industry)
Responsible Party: Principal Investigator, RAQUEL ESCALERA, MD, Surgery Department., Hospital del SAS de Jerez
Other Study IDs: SLN_GC_SPIO_RE_18
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer (GC); Sentinel Lymph Node Biopsy (SLNB)
Keywords: GASTRIC CANCER, SENTINEL LYMPH NODE, OSNA, DUAL TRACER
MeSH Terms: conditions — Stomach Neoplasms | interventions — ferric oxide; Methylene Blue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS WITH GASTRIC CANCER AND CK19+
  Interventions: Procedure: Dual tracer: The infiltration of the Supermagnetic Iron Oxide (SPIO) and Methylene Blue; Diagnostic Test: OSNA AND H-E

INTERVENTIONS:
Procedure: Dual tracer: The infiltration of the Supermagnetic Iron Oxide (SPIO) and Methylene Blue — Participation in the study did not alter the indications or standard surgical technique. The only additional intervention consisted of intraoperative administration of SPIO, performed either laparoscopically or conventionally, as appropriate.
  Immediately after removal of the surgical specimen : Submucosal instillation of methylene blue was then performed at the tumour periphery
Diagnostic Test: OSNA AND H-E — Analysed the performance of one-step nucleic acid amplification (OSNA) versus conventional histology and applied pooling analysis with OSNA in non-sentinel nodes

SUMMARY:
Gastric cancer (GC) remains an oncological challenge, where lymph node involvement is a key prognostic factor. Sentinel lymph node (SLN) mapping may improve staging and reduce surgical morbidity. This study evaluated a dual-tracer technique - superparamagnetic iron oxide (SPIO) and methylene blue - for ex vivo SLN detection in GC, analysed the performance of one-step nucleic acid amplification (OSNA) versus conventional histology and applied pooling analysis with OSNA in non-sentinel nodes.

The aim of this prospective study was, firstly, to evaluate the accuracy of ex vivo SLN detection using a novel dual tracer: SPIO not previously used for this pathology, combined with methylene blue. Secondly, to perform a diagnostic concordance analysis between the results of the conventional histological haematoxylin-eosin (H-E) study versus the OSNA (One Step Nucleic Acid Amplification) molecular method, for the detection of lymph node metastases in patients with gastric cancer undergoing surgery with curative intent and lymphadenectomy.

DETAILED DESCRIPTION:
Observational, prospective and analytical study, carried out in a second level university hospital with 500 inpatient beds.

All patients with an indication for oncological gastric surgery who met the inclusion criteria were consecutively included in the period between August 2017 and March 2022.

All patients were diagnosed, treated and followed up according to the centre's standard clinical practice, following a protocol based on the scientific evidence collected in the European ESMO-ESSO-ESTRO guidelines for the management of gastric cancer Surgical procedures Participation in the study did not alter the indications or standard surgical technique. The only additional intervention consisted of intraoperative administration of SPIO (superparamagetic iron oxide)

Variables collected For each patient included in the study, demographic, clinical and pathological variables were systematically collected: age, sex, type of neoplasm, size, tumour grade, TNM 8ed, stage, neoadjuvant treatment and degree of regression, if any. Perioperative variables such as type of intervention, type of lymphadenectomy, time of infiltration and tracer detection, operative complications, reoperation rate and hospital stay were also evaluated. During follow-up, oncological variables such as recurrence rate, mortality, overall survival and disease-free survival were analysed.

Statistical analysis Data were analysed using SPSS version 26.0 software (IBM Corp., Armonk, NY, USA) and EpiDat version 4.2 (Xunta de Galicia, Spain). A descriptive analysis was performed using measures of central tendency and dispersion for quantitative variables, and absolute and relative frequencies for qualitative variables. The chi-square test with correction was used to compare qualitative variables. Concordance between methods was assessed using Cohen's kappa coefficient. Diagnostic accuracy was determined by calculating sensitivity and specificity, together with their respective 95% confidence intervals according to Hanley&McNeil. Survival curves were estimated using the Kaplan-Meier method, and differences between groups were analysed using the log-rank test. A value of p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a diagnosis of gastric adenocarcinoma, undergoing surgery with curative intent by total or subtotal gastrectomy, accompanied by D1, D1+ or D2 lymphadenectomy, and with preoperative positivity for cytokeratin 19 (CK19) in the tumour sample.

Exclusion Criteria:

* Patients with gastric cancer recurrence, those diagnosed with other active neoplasms, metastatic disease at diagnosis, as well as patients with Siewert type I and II gastrooesophageal junction carcinoma. Neoadjuvant treatment was not considered an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an indication for oncological gastric surgery who met the inclusion criteria were consecutively included in the period between August 2017 and March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
demographic, clinical and pathological variables | cut-off date for all patients: 15 July 2025.
  For each patient included in the study, demographic, clinical and pathological variables were systematically collected: age, sex, type of neoplasm, size, tumour grade, TNM 8ed, stage, neoadjuvant treatment and degree of regression, if any. Perioperative variables such as type of intervention, type of lymphadenectomy, time of infiltration and tracer detection, operative complications, reoperation rate and hospital stay were also evaluated. During follow-up, oncological variables such as recurrence rate, mortality, overall survival and disease-free survival were analysed

SECONDARY OUTCOMES:
Migration times of both tracers | Immediately after surgery
  the SLNs stained with methylene blue and/or those detected using the Sentimag® probe, previously calibrated, were dissected and extracted
Lymph node involvement | 6 MONTHS
  Each lymph node identified, including the sentinels obtained in the operating theatre, was sectioned into two symmetrical halves: one for conventional histopathological analysis and the other for molecular analysis by OSNA

CONTACTS AND LOCATIONS:
Overall Officials: ESCALERA-PEREZ, RAQUEL, MD, Principal Investigator — Hospital del SAS de Jerez
Locations (1):
- Univesrsity Hospital of Jerez Frontera, Jerez de la Frontera, CADIZ, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known whether there will be a plan for the IPD to be made available